CLINICAL TRIAL: NCT05777798
Title: Multicentric Clinical Investigation on the Use of Single-dose Ophthalmic Solution Based on Hyaluronate Sodium Phosphate in the Treatment of Eye Discomfort in Particular in Case of Ocular Dryness
Brief Title: Clinical Investigation on the Use of Ophthalmic Solution Based on Sodium Hyaluronate in Treatment of Eye Discomfort
Status: Completed | Type: Observational
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: 052/SI Hyalistil Bio PF Mono
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Ocular Dryness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hyalistil Bio PF — Moisturizing and lubricating ophthalmic solution

SUMMARY:
The purpose of this study is to assess the performance and safety resulting from the treatment of an ophthalmic solution for the ocular discomfort and in particular in presence of ocular dryness.

DETAILED DESCRIPTION:
Multicenter, prospective, observational, open-label, non- interventional clinical investigation evaluating the performance and safety of 4 daily instillations of the ophthalmic solution in the treatment of mild irritation of the ocular surface.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (male or female) must be ≥ 18 years of age;
2. Subject able to provide Informed Consent, in compliance with the good clinical practice and local laws (thus, subject able to comprehend the full nature and purpose of the study, including possible risks and side effects);
3. Subjects with ocular discomfort resulting from mild to moderate dry eye in one or both eyes determined by:

   * Scoring of ocular surface staining with fluorescein using the National Eye Institute (NEI) scale. Total score per single eye range 6-33 summing the score of cornea and conjunctiva. (Considering a normal score of 0-33);
   * Tear film break-up time with fluorescein (TFBUT) ≤ 10 seconds; The TFBUT value will be recorded as the average of 3 measurements;
   * Symptom Assessment in Dry Eye (SANDE) questionnaire ≥ 35.
4. Subject able to be compliant with the requirements of the clinical investigation plan, according to the Investigator;
5. Subject who qualifies for Hyalistil Bio PF treatment according to the approved indication;
6. Subject who in physician's opinion will benefit from this treatment.

Exclusion Criteria:

1. Corneal injuries or abrasions of traumatic origin in the eye of study;
2. Ocular infection or clinically significant inflammation (such as Herpes Simplex infection, corneal virus infection, bacterial, viral or fungal conjunctivitis, tuberculosis and mycosis of the eye, purulent and herpetic blepharitis, stye);
3. Sjögren's syndrome;
4. Stevens-Johnson syndrome;
5. Systemic lupus erythematosus;
6. Pathologies associated with corneal thinning;
7. Taking drugs that may interfere with tear gland secretion (beta -blockers);
8. Patients using any topical therapies such as non-steroidal antiinflammatory drugs, cortisone, cyclosporine, vasoconstrictor, artificial tears (different than the investigated product) the eye of study;
9. Treatment with topical or systemic corticosteroids in the 4 weeks preceding the study;
10. Known or potential hypersensitivity and/or history of allergic reactions to one of the components of the topical medical device.
11. Participation in another clinical trial within the previous 30 days;
12. Evidence of severe or uncontrolled systemic disease or any other significant disorders, which in the opinion of the Investigator does not allow the participation in the study or could compromise the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 28 male and female subjects with signs and symptoms of ocular discomfort and ocular irritation resulting from ocular dryness who qualifies for Hyalistil Bio PF treatment.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Scollo, M.D., Principal Investigator — U.O.S. Oculistica "San Marco" A.O.U. Policlinico "G.Rodolico-San Marco" Catania, Italy
Locations (2):
- Italy (2):
  - P.O. San Marco, Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco" Oculistica,, Catania, CT
  - U.O. di Oculistica, Presidio Belmonte, Azienda Ospedaliero Universitaria Policlinico "Paolo Giaccone", Palermo

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with signs and symptoms of ocular discomfort and ocular irritation resulting from ocular dryness / tear film alterations
Units Other Than Participants: one eye (the worst eye)
Groups:
- Hyalistil Bio PF: 28 subjects were treated for 30 days with 4 daily instillations of Hyalistil Bio PF.
Period: Overall Study
Arm/Group | Hyalistil Bio PF
Started | 28; 28 one eye (the worst eye)
Completed | 28; 28 one eye (the worst eye)
Not Completed | 0; 0 one eye (the worst eye)

BASELINE CHARACTERISTICS:
Units Other Than Participants: worst eye
Groups:
- Hyalistil Bio PF: 28 male and female subjects with signs and symptoms of ocular discomfort were treated for 30 days with 4 daily instillations of Hyalistil Bio PF.
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
Number analyzed (worst eye) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.46 (55.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 28
TFBUT (Tear Film Break Up Time) [Mean (Standard Deviation); unit: Second] — The TFBUT has been performed after instillation of 5 microliters of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. The patient was instructed to blink several times to mix the fluorescein with the tear film. To achieve maximum fluorescence, before evaluating TFBUT, the examiner waited approximately 30 seconds after instillation . The TFBUT was measured by determining the time to tear break-up within 10 seconds during the first minute after the instillation of the fluorescein.
  Second | 5 (2.03)

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Break-up Time With Fluorescein (TFBUT)
Description: The TFBUT will be performed after instillation of 5 microliters of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. The patient will be instructed to blink several times to thoroughly mix the fluorescein with the tear film. To achieve maximum fluorescence, the examiner should wait approximately 30 seconds after instillation before evaluating TFBUT. The TFBUT was measured by determining the time in seconds to tear break-up within 10 seconds maximum, and it was measured three time during the first minute after the instillation of fluorescein solution. The TFBUT value will be the average of 3 measurements.
Time Frame: Evaluated at Visit 1 (baseline) and Visit 3 (day 35 ± 4 - study termination)
Population: A total of 28 patients were screened and included in the FAS (ITT analysis) and in the Safety population. Three out of 28 patients had a major protocol deviation, one patient did not show up for the study termination visit, two patients did not meet the exclusion criteria "Taking drugs that may interfere with tear gland secretion (beta -blockers)". Thus, the PP population consisted of 25 patients.
Measure: Mean (Standard Deviation); unit: Second
Units Other Than Participants: the worst eye
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
Number analyzed (the worst eye) | 28
Second
  TFBUT at Visit 1 (Baseline) | 5.00 (2.03)
  TFBUT at Visit 3 (Study termination): number analyzed (Participants) | 25
  TFBUT at Visit 3 (Study termination): number analyzed (the worst eye) | 25
  TFBUT at Visit 3 (Study termination) | 13.46 (5.83)

2. Secondary Outcome: Fluorescein Staining
Description: The NEI/Industry Workshop scale (1995) is an ophthalmological rating scale developed by the National Eye Institute (NEI, USA) to measure the degree of corneal and conjunctival staining after instillation of fluorescein or rose bengal/lissamine green.
  * The cornea is divided into 5 zones: Central, Superior, Inferior, Nasal, Temporal. Each zone is assigned a score from 0 to 3: 0 = no staining; 1 = mild; 2 = moderate; 3 = severe (Lower values=better outcomes - Total maximum cornea staining = 15).
  * The bulbar conjunctiva is divided into 6 areas: Superior nasal, Inferior nasal, Superior temporal, Inferior temporal, Superior (under the upper eyelid, less frequently assessed), Inferior (above the inferior fornix). The total maximum conjunctiva staing is 18.
  The total staining score is given by the sum of the corneal and conjunctival staining (Lower values=better outcomes - Min=0, Max=33).
Time Frame: Evaluated at Visit 1 (baseline), Visit 2 (day 14± 2) and Visit3 (day 35 ± 4 - study termination visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
score on a scale
  Total NEI Score at Visit 1 (baseline) | 16.82 (5.48)
  Total NEI Score at Visit 2 | 9.79 (3.45)
  Total NEI Score at Visit 3 (Study Termination Visit) | 5.18 (2.46)

3. Secondary Outcome: SANDE
Description: The SANDE questionnaire (Symptom Assessment in Dry Eye) is a very simple, validated tool to assess dry eye symptoms.
  It's based on two visual analog scale (VAS) questions that measure: 1) Frequency of symptoms (dry and irritated); 2) Severity of symptoms (dryness and irritation).
  Each question is scored by the patients on a 0-100 mm VAS line (0 = no symptoms, 100 = maximum symptoms), marking the point that they feel represents their perception of their current state.
  Data collected from the SANDE questionnaire were calculated by multiplying the frequency score by the severity score and obtaining the square root.
Time Frame: Evaluated at Visit 1 (baseline), Visit2 (day 14± 2) and Visit3 (35 ± 4 - study termination)
Measure: Mean (Standard Deviation); unit: score on scale (millimeters)
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
score on scale (millimeters)
  Total score severity: Visit 1 (baseline) | 67.32 (16.53)
  Total score severity: Study termination | 26.43 (22.15)
  Total score frequency: Visit 1 (baseline) | 67.68 (17.08)
  Total score frequency: Study termination | 27.14 (25.07)

4. Secondary Outcome: Evaluation of the Degree of Satisfaction to the Treatment Reported by Patients Through the Use of the Visual Analogue Scale (VAS).
Description: To evaluate the degree of satisfaction of patients to the treatment we used the visual analogue scale (VAS) ranging from 0 to 100 mm in a horizontal line.
  Patients will be asked to place a vertical mark (on the horizontal line, from 0 to100 mm) to indicate the degree of satisfaction to the treatment, where: 0-10 mm=no: 1-30 mm=very mild; 31-50 mm=mild; 51-70 mm=moderate; 71-90 mm=strong; 91-100 mm=very strong.
  Patients were asked to rate their level of satisfaction answering each of these questions: 1) "I feel satisfied using this treatment? ''; 2) "With this treatment, I have a feeling of freshness?"; 3) "With this treatment, I have a feeling of relief?"; 4) "This treatment contributed to reduce my pain due to eye dryness?''; 5) "This treatment is comfortable? '' The response results are expressed in frequency and percentage of the total for each of the questions in the categories "very mild", "mild", "moderate", "strong" and "very strong".
Time Frame: Evaluated at day 35 ± 4 of treatment
Population: Frequency missing = 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 27
Participants
  1) "I feel satisfied using this treatment?": very mild | 0
  1) "I feel satisfied using this treatment?": mild | 4
  1) "I feel satisfied using this treatment?": moderate | 3
  1) "I feel satisfied using this treatment?": strong | 12
  1) "I feel satisfied using this treatment?": very strong | 8
  2) "With this treatment, I have a feeling of freshness?": very mild | 2
  2) "With this treatment, I have a feeling of freshness?": mild | 1
  2) "With this treatment, I have a feeling of freshness?": moderate | 3
  2) "With this treatment, I have a feeling of freshness?": strong | 14
  2) "With this treatment, I have a feeling of freshness?": very strong | 7
  3) "With this treatment, I have a feeling of relief?": very mild | 1
  3) "With this treatment, I have a feeling of relief?": mild | 2
  3) "With this treatment, I have a feeling of relief?": moderate | 2
  3) "With this treatment, I have a feeling of relief?": strong | 15
  3) "With this treatment, I have a feeling of relief?": very strong | 7
  4) "This treatment contributed to reduce my pain due to eye dryness?'': very mild | 0
  4) "This treatment contributed to reduce my pain due to eye dryness?'': mild | 2
  4) "This treatment contributed to reduce my pain due to eye dryness?'': moderate | 4
  4) "This treatment contributed to reduce my pain due to eye dryness?'': strong | 14
  4) "This treatment contributed to reduce my pain due to eye dryness?'': very strong | 7
  5) "This treatment is comfortable? '': very mild | 0
  5) "This treatment is comfortable? '': mild | 2
  5) "This treatment is comfortable? '': moderate | 2
  5) "This treatment is comfortable? '': strong | 11
  5) "This treatment is comfortable? '': very strong | 12

5. Secondary Outcome: Dry Eye-Related Quality of Life (DEQS Total Score)
Description: Quality of life was assessed using the Dry Eye-Related Quality of Life Score (DEQS) questionnaire, which includes 15 items grouped into two subscales: Symptom Burden (6 items) and Impact on Daily Life (9 items). Each item is scored on a 0 to 4 scale, with higher scores indicating worse symptoms. Subscale scores range from 0 to 24 and 0 to 36, respectively. A total DEQS score was calculated by summing all item scores and converting the raw total to a 0-100 scale, where lower scores indicate better quality of life.
Time Frame: Baseline (Visit 1) and Study Termination Visit (Day 35 ± 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
score on a scale
  DEQS Summary score - Visit 1 baseline | 53.87 (13.44)
  DEQS Summary score - Study Termination V | 24.08 (17.13)
  DEQS Bothersome Ocular Symptoms subscale Visit 1 baseline | 56.37 (13.72)
  DEQS Bothersome Ocular Symptoms subscale Study Termination Visit | 23.25 (16.70)
  DEQS Impact on Daily Life subscale Visit 1 baseline | 51.96 (17.26)
  DEQS Impact on Daily Life subscale Study Termination Visit | 23.81 (19.31)

6. Secondary Outcome: Tear Film Break-up Time With Fluorescein (TFBUT)
Description: as for outcome 1
Time Frame: Evaluated at day 14 ± 2 of treatment (Visit 2) and day 35 ± 4 of treatment (Visit 3 - Study termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Second
Units Other Than Participants: the worst eye
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
Number analyzed (the worst eye) | 28
Second
  TFBUT at Visit 2: number analyzed (Participants) | 26
  TFBUT at Visit 2: number analyzed (the worst eye) | 26
  TFBUT at Visit 2 | 10.27 (5.01)
  TFBUT at Visit 3 (Study termination): number analyzed (Participants) | 25
  TFBUT at Visit 3 (Study termination): number analyzed (the worst eye) | 25
  TFBUT at Visit 3 (Study termination) | 13.46 (5.83)

7. Secondary Outcome: Best Corrected Visual Acuity (BCVA)
Description: The ETDRS chart uses a standardized, logarithmic letter chart (Sloan letters, 5 per line). Results can be reported as either logMAR values or letter scores, in our study we used the "Line method" (the smallest line where at least 3 of 5 letters are correctly read), while Visual Acuity was expressed as Snellen Distance Equivalent (meters); in the Italian decimal system, 10/10 corresponds to 6/6" or 0.0 logMAR.
  To maintain consistency across clinics and trials, the examination conditions were standardized as follow: Test distance 4 meters, Chart uniformly illuminated (~85 cd/m² luminance), with a white, high contrast (≥ 90%) background, the Best corrected visual acuity (BCVA) was measured with trial frame lenses.
  The BCVA was testing monocularly, while the patient was encouraged to read as many letters as possible, even if guessing.
  When the patient misses a prespecified number (3 or more errors in a row), testing stops.
Time Frame: Evaluated at day 14± 2 and 35 ± 4 of treatment versus baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
Participants
  BCVA Visit 1 (Baseline): BCVA = 0.6/10 (logMAR 1.2) | 1
  BCVA Visit 1 (Baseline): BCVA = 6/10 (logMAR 0.2) | 2
  BCVA Visit 1 (Baseline): BCVA = 9/10 (logMAR 0.05) | 2
  BCVA Visit 1 (Baseline): BCVA = 10/10 (logMAR 0.0) | 23
  BCVA Visit 2: BCVA = 0.6/10 (logMAR 1.2) | 1
  BCVA Visit 2: BCVA = 6/10 (logMAR 0.2) | 2
  BCVA Visit 2: BCVA = 9/10 (logMAR 0.05) | 2
  BCVA Visit 2: BCVA = 10/10 (logMAR 0.0) | 23
  BCVA Study Termination Visit: BCVA = 0.6/10 (logMAR 1.2) | 1
  BCVA Study Termination Visit: BCVA = 6/10 (logMAR 0.2) | 2
  BCVA Study Termination Visit: BCVA = 9/10 (logMAR 0.05) | 1
  BCVA Study Termination Visit: BCVA = 10/10 (logMAR 0.0) | 24

8. Other Pre Specified Outcome: Investigator Global Assessment of Safety (IGAS)
Description: Safety was assessed using the Investigator Global Assessment of Safety (IGAS), a 4-point categorical scale where 1 = very good safety, 2 = good safety, 3 = moderate safety, and 4 = poor safety. IGAS was evaluated at the Study Termination Visit and summarized by reporting the number and percentage of participants in each category.
Time Frame: Study Termination Visit (Day 35 ± 4)
Population: One patient did not show up to study termination visit
Measure: Count of Participants; unit: Participants
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 27
Participants
  Point scale 1 (very good safety) | 27
  Point scale 2 (good safety) | 0
  Point scale 3 (moderate safety) | 0
  Point scale 4 (poor safety) | 0

9. Other Pre Specified Outcome: Change in Intraocular Pressure (IOP)
Description: Intraocular pressure (IOP) was measured in mmHg using Goldmann applanation tonometry after topical anesthesia with unpreserved 0.4 percent oxybuprocaine hydrochloride. IOP was assessed at three pre-specified study visits: baseline (Visit 1), Visit 2 during treatment, and the Study Termination Visit. Results were summarized by visit for all participants included in the intention-to-treat population.
Time Frame: Baseline (Visit 1), Visit 2 (Day 14 ± 2), and Study Termination Visit (Day 35 ± 4)
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Groups:
- Hyalistil Bio PF: 28 male and female subjects with signs and symptoms of ocular discomfor were treated for 30 days with 4 daily instillations of Hyalistil Bio PF.
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
millimeters of mercury
  IOP - Visit 1 | 12.86 (2.00)
  IOP - Visit 2 | 12.82 (1.44)
  IOP - Visit 3 Study termination Visit | 12.61 (1.32)

10. Other Pre Specified Outcome: Treatment Compliance Rate
Description: Treatment compliance was assessed during the treatment period by counting returned single-dose containers and boxes at the Study Termination Visit. Compliance was calculated as the percentage of prescribed doses administered relative to planned doses for each participant. Participants were categorized into predefined compliance categories (<50%, 50-80%, >80%) for reporting purposes.
Time Frame: During the treatment period, assessed at Study Termination Visit (Day 35 ± 4)
Measure: Count of Participants; unit: Participants
Arm/Group | Hyalistil Bio PF
Number analyzed (Participants) | 28
Participants
  < 50% = Poor Compliance | 1
  50-80% = Moderate Compliance | 2
  > 80% = Good Compliance | 25

ADVERSE EVENTS:
Time Frame: The period of time that Adverse Event (AEs) data were collected for a maximum of 37 days. The Time Frame for all participant was from enrollment until end of follow-up. Specifically, for the ITT population (days/number of participants): 14/1 (missing), 33/7, 34/11, 35/6, 36/1, 37/2; for PP population (days/number of participants): 32/1, 33/7, 34/9, 35/5, 36/1 and 37/2.
Description: All adverse event/incidents/potentially incidents (independently from the seriousness) experienced during the study, spontaneously reported by the patient, or elicited as a result of general questioning by the site staff, were recorded in the source documents (Clinical Record) and on the eCRF. No Adverse Events were collected in the source documents (Medical Record) and in the eCRF that are not reported here.
Arm/Group | Hyalistil Bio PF
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT05777798/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT05777798/SAP_001.pdf